CLINICAL TRIAL: NCT01955109
Title: Open-label Follow-up Study of the VIPES Study to Evaluate Long-term Efficacy and Safety of the Viaskin Peanut
Brief Title: Follow-up of the VIPES Study to Evaluate Efficacy and Safety of Viaskin Peanut in Adults and Children
Acronym: OLFUS-VIPES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DBV Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLFUS-VIPES; 2013-001754-10 (EudraCT Number)
Record Dates: First submitted 2013-09-24; First posted 2013-10-07 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Peanut Allergy
Keywords: Food allergy; Immediate hypersensitivity; Whole peanut extract; Allergenic product; Specific Immunotherapy; Epicutaneous Immunotherapy (EPIT)
MeSH Terms: conditions — Peanut Hypersensitivity; Food Hypersensitivity; Hypersensitivity, Immediate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Viaskin Peanut 250 mcg (Experimental)
  Interventions: Biological: Viaskin Peanut 250 mcg

INTERVENTIONS:
Biological: Viaskin Peanut 250 mcg — Subjects epicutaneously administered for 24 hours every 24 hours with a patch containing 250 mcg peanut proteins as whole peanut extract

SUMMARY:
The objectives of this open-label follow-up study for subjects who previously were randomized and have completed the VIPES study for the treatment of peanut allergy, are:

* To assess the efficacy of Viaskin Peanut after up to 36 months of treatment.
* To evaluate the safety of long-term treatment with Viaskin Peanut.
* To evaluate sustained unresponsiveness to peanut after a period of 2 months without treatment in subjects showing desensitization to peanut after treatment with Viaskin Peanut.

DETAILED DESCRIPTION:
Peanut allergy is a common allergy in the United States, with a prevalence in the general population as high as 1%. Peanut allergy management is based on strict peanut avoidance and injectable epinephrine after the allergic systemic reactions have started. Specific Immunotherapy methods currently available have shown some limitations in their use because of safety issues. Hence, there is an important unmet medical need for efficient and safe treatment of peanut allergy.

DBV Technologies has developed an epicutaneous delivery system, called Viaskin, a method based on delivering precise quantity of the allergen on the upper layers of the skin. Avoiding contact between the allergen and the bloodstream should confer to epicutaneous immunotherapy (EPIT) a higher level of safety as systemic reactions should be circumvented

The OLFUS-VIPES study is an open-label follow-up study for subjects who previously were randomized and have completed the VIPES efficacy and safety study. Subjects will be offered enrollment in this follow-up study to receive an additional 24 months of Viaskin Peanut treatment followed by a period of 2 months without treatment while maintaining a peanut-free diet.

The trial will be conducted at the same sites as the VIPES study with investigators and staff trained and experienced in the diagnosis and the management of peanut allergy and anaphylaxis, and who are capable of performing a double-blind placebo-controlled food challenge (DBPCFC) in adult and/or pediatric subjects.

According to the current amended study protocol, all subjects enrolling into the OLFUS-VIPES study after having completed the VIPES study will receive the highest dose of Viaskin Peanut, i.e. 250 mcg peanut protein, regardless of prior treatment (placebo, 50 mcg, 100 mcg or 250 mcg Viaskin Peanut) they were receiving in the VIPES study. Subjects who already enrolled into the OLFUS-VIPES study under the initial protocol design will all switch to receive the 250 mcg dose at Month 6 or at Month 12 of treatment in the OLFUS-VIPES study upon approval of the amended protocol at their sites. The study will remain blinded for all subjects until the VIPES study is unblinded. All subjects completing the OLFUS-VIPES study should receive overall 24 months of active treatment followed by a period of 2 months without treatment for those subjects being assessed for sustained unresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric subjects (≥7 years) who completed the VIPES study, with a mandatory and documented DBPCFC at Month 12 in the VIPES study.
* Signed informed consent from adult subjects or parent(s)/guardian(s) of children <18 years and children's assent for children >7 years or as per country-specific regulations or laws. This consent should be signed no later than Visit 11 in the VIPES study.
* Negative pregnancy test for women of childbearing potential at Visit 10 in the VIPES study.
* Female subject of childbearing potential must use effective methods of contraception to prevent pregnancy and agree to continue to practice an acceptable method of contraception for the duration of participation in the study. Documented sexual abstinence will be accepted as an effective method of contraception for girls below 15 years of age.
* Subjects and/or parents/guardians willing to comply with all study requirements during their participation in the study.

Exclusion Criteria:

* Severe reaction during the DBPCFC at Month 12 in the VIPES study, defined as need for intubation, hypotension persisting after epinephrine administration, and/or the need for more than two doses of epinephrine.
* Pregnancy or lactation.
* Females of childbearing potential planning a pregnancy in the coming 2 to 3 years.
* Subjects who became allergic to chocolate or who do not want to consume the chocolate study challenge vehicle anymore.
* Subjects who developed hypersensitivity to excipients of the Viaskin patches or of the food challenge formula used during the VIPES study.
* Inability to discontinue short-acting antihistamines for three days or long-acting antihistamines for five to seven days (depending on half-life) prior to skin prick testing or food challenges.
* Subjects with asthma that has evolved and now fulfills any of the criteria defined as follows:

  * uncontrolled persistent asthma by National Asthma Education and Prevention Program Asthma guidelines (2007) or by Global Initiative for Asthma (2011) or being treated with combination therapy of medium dose inhaled corticosteroid with a long acting inhaled β2-agonists.
  * at least two systemic corticosteroid courses for asthma in the past year or one oral corticosteroid course for asthma in the past three months.
  * prior intubation for asthma in the past year.
* Subjects receiving β-blocking agents, angiotensin-converting enzyme inhibitors, angiotensin-receptor blockers, calcium channel blockers or tricyclic antidepressant therapy.
* Subjects receiving or planning to receive anti-tumor necrosis factor drugs or anti-IgE drugs (such as omalizumab) or any biologic immunomodulatory therapy.
* Subjects receiving or planning to receive any type of immunotherapy to any food (e.g. oral immunotherapy, sublingual immunotherapy, specific oral tolerance induction) during their participation in the study.
* Subjects receiving or planning to receive any aeroallergen immunotherapy during their participation in the study.
* Allergy or known history of reaction to Tegaderm® with no possibilities to use an alternative dressing approved by the sponsor.
* Subjects suffering from generalized dermatologic disease (e.g. severe atopic dermatitis, uncontrolled generalized eczema, ichthyosis vulgaris) with no intact zones to apply the patches.
* Any new disorder in which epinephrine is contraindicated such as coronary artery disease, uncontrolled hypertension, or serious ventricular arrhythmias.
* A history of non compliance in the VIPES study. Non compliance is defined as subjects not applying the patch at all for 60 days or more (this can be either consecutive or intermittent non-application of the patches) during the whole VIPES study duration
* Participation in another clinical intervention study in the past year, other than the VIPES study.
* Subjects on any experimental drugs in the past year, other than those used in the VIPES study.

Other inclusion/exclusion criteria may apply.

Ages: 7 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 171 (Actual)
Dates: Start 2013-09; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (10):
  - University of California, Rady Childrens Hospital, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Childrens' Hospital, Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
  - ASTHMA, Inc., Seattle, Washington
- Canada (4):
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Asthma Research Institute, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario
  - Centre de Recherche Appliquée en Asthme et Allergie de Québec, Sainte-Foy, Quebec
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux, Hôpital Pellegrin, Bordeaux
  - Hôpital Saint Vincent de Paul, Lille
  - GCS des hôpitaux pédiatriques, Nice
  - Hôpital Necker, Paris
  - Nouvel Hôpital Civil, Strasbourg
  - Hôpitaux De Brabois, Vandœuvre-lès-Nancy
- Netherlands (2):
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht

REFERENCES:
- [Derived] Lewis MO, Brown-Whitehorn TF, Cianferoni A, Rooney C, Spergel JM. Peanut-allergic patient experiences after epicutaneous immunotherapy: peanut consumption and impact on QoL. Ann Allergy Asthma Immunol. 2019 Jul;123(1):101-103. doi: 10.1016/j.anai.2019.04.006. Epub 2019 Apr 10. No abstract available. PMID 30978404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children, adolescent and adult participants who were previously randomized in and completed the VIPES study (V712-202; NCT01675882) were eligible to enroll in this Phase II open-label follow-up study to receive an additional 24 months of Viaskin® Peanut (DBV712) Epicutaneous Immunotherapy (EPIT). Participants were enrolled in 21 study centers in 4 countries in France, the Netherlands, Canada and the USA from 30 August 2013 and the last participant completed 29 September 2016.
Pre-assignment Details: Participants who received 50, 100 or 250 micrograms (μg) Viaskin Peanut in VIPES continued on same dose in OLFUS-VIPES; those receiving placebo were re-randomized 1:1:1 to 50, 100 or 250 μg Viaskin Peanut. After protocol amendment 1, all participants received 250 μg dose from start of OLFUS-VIPES; those already enrolled were switched to 250 μg at Month 6 visit.
Groups:
- VIPES Initial Treatment Group: All Viaskin Peanut Doses: Participants were randomized in the VIPES study to receive either 50 μg, 100 μg or 250 μg Viaskin Peanut for 12 months. In the follow-up OLFUS-VIPES study, participants received 250 μg Viaskin Peanut for up to 24 months. Participants received treatment with Viaskin Peanut for a total of up to 36 months.
- VIPES Initial Treatment Group: Placebo: Participants were randomized in the VIPES study to receive placebo for 12 months. In the follow-up OLFUS-VIPES study, participants received 250 μg Viaskin Peanut for up to 24 months. Participants received treatment with Viaskin Peanut for a total of up to 24 months.
Period: Overall Study
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Started | 123 | 48
Completed Study Until Month 12 | 103 | 46
Completed (Completed Month 24 (or Month 26 if applicable)) | 78 | 39
Not Completed | 45 | 9
Not completed — Adverse Event | 2 | 0
Not completed — Participant unwilling to continue | 35 | 7
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Non-compliance | 3 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who received at least 1 dose of investigational product (IP) during the OLFUS-VIPES study.
Groups:
- Total: Total of all reporting groups
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo | Total
Number analyzed (Participants) | 123 | 48 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age at OLFUS-VIPES entry.
  years | 13.7 (6.64) | 13.0 (6.59) | 13.5 (6.61)
Age, Customized [Count of Participants; unit: Participants] — Participants' ages at OLFUS-VIPES entry.
  Participants
    Children (6-11 years) | 60 | 23 | 83
    Adolescents (12-17 years) | 34 | 18 | 52
    Adults (18-55 years) | 29 | 7 | 36
    Adolescents and Adults (12-55 years) | 63 | 25 | 88
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 18 | 61
  Male | 80 | 30 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The ethnicity of the participants at French local sites was not collected as it was not applicable as per local law. As such, these participants are included in the category of 'Not applicable'
  Participants
    Caucasian | 80 | 28 | 108
    Black | 3 | 2 | 5
    Hispanic | 1 | 2 | 3
    Asian | 16 | 4 | 20
    Other | 5 | 3 | 8
    Not applicable | 18 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Canada | 40 | 14 | 54
  Netherlands | 5 | 1 | 6
  United States | 60 | 24 | 84
  France | 18 | 9 | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment Responders at Months 12 and 24
Description: A treatment responder was defined as a participant with a peanut protein eliciting dose (ED) equal to or greater than 1000 milligram (mg) peanut protein or with at least a 10-fold increase of the ED compared to their initial ED observed at the VIPES baseline, as determined by double-blind placebo-controlled food challenge (DBPCFC) at Months 12 and 24. At Month 12, participants had received 24 months of active treatment for those who received Viaskin Peanut in the VIPES study, and 12 months of active treatment for those who received placebo in the VIPES study. At Month 24, participants had received 36 months of active treatment for those who received Viaskin Peanut in the VIPES study, and 24 months of active treatment for those who received placebo in the VIPES study. The percentage of responders at Month 12 and Month 24 are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: Month 12 and Month 24 (end of treatment) of the OLFUS-VIPES study
Population: The full analysis set was the intent-to-treat population which consisted of all participants and results are reported for those participants who had the Months 12 and 24 DBPCFC performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 123 | 48
percentage of participants
  Month 12: number analyzed (Participants) | 103 | 46
  Month 12 | 64.1 [54.0 to 73.3] | 50.0 [34.9 to 65.1]
  Month 24: number analyzed (Participants) | 83 | 41
  Month 24 | 67.5 [56.3 to 77.4] | 58.5 [42.1 to 73.7]

2. Secondary Outcome: Percentage of Participants Unresponsive to a Cumulative Dose of at Least 1440 mg Peanut Protein at Month 24
Description: Participants were considered unresponsive if they showed no objective symptoms leading to stopping the challenge during the Month 24 DBPCFC with a cumulative dose of at least 1440 mg of peanut protein, up to a cumulative dose of 5044 mg peanut protein. The percentage of unresponsive participants is presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: Month 24 (end of treatment) of the OLFUS-VIPES study
Population: The full analysis set was the intent-to-treat population which consisted of all participants and results are reported for those participants who had the Month 24 DBPCFC performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 83 | 41
percentage of participants | 31.3 [21.6 to 42.4] | 7.3 [1.5 to 19.9]

3. Secondary Outcome: Percentage of Participants With a Sustained Unresponsiveness to a Cumulative Dose of at Least 1440 mg Peanut Protein at Month 26
Description: Participants who were unresponsive to a cumulative dose of 1440 mg of peanut protein or above at the Month 24 DBPCFC, had an additional 2-month period without treatment and continued on a peanut-free diet to assess for sustained unresponsiveness by a DBPCFC at Month 26. The percentage of participants with this sustained unresponsiveness, i.e, who showed no objective symptoms leading to stopping the challenge during the DBPCFC to a cumulative dose of 1440 mg of peanut protein or above at Month 26, are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: Month 26 (2 months post-treatment) of the OLFUS-VIPES study
Population: The full analysis set was the intent-to-treat population which consisted of all participants and results are reported for participants who had the Month 26 DBPCFC performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 22 | 3
percentage of participants | 77.3 [54.6 to 92.2] | 100 [29.2 to 100.0]

4. Secondary Outcome: Median Cumulative Reactive Dose of Peanut Protein at Months 12 and 24
Description: The cumulative reactive dose was defined as the sum of all peanut protein doses taken by the participant during the DBPCFC. To distinguish participants who reached the highest dose of the DBPCFC without objective symptoms 1000 mg was added to the cumulative reactive dose to obtain an adjusted value. The median cumulative reactive doses at Months 12 and 24 are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: Month 12 and Month 24 (end of treatment) of the OLFUS-VIPES study
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 123 | 48
mg
  Month 12: number analyzed (Participants) | 103 | 46
  Month 12 | 480.0 [140.0 to 2240.0] | 365.0 [140.0 to 1440.0]
  Month 24: number analyzed (Participants) | 83 | 41
  Month 24 | 440.0 [160.0 to 3040.0] | 440.0 [140.0 to 1440.0]

5. Secondary Outcome: Mean Cumulative Reactive Dose of Peanut Protein at Months 12 and 24
Description: The cumulative reactive dose was defined as the sum of all peanut protein doses taken by the participant during the DBPCFC. To distinguish participants who reached the highest dose of the DBPCFC without objective symptoms 1000 mg was added to the cumulative reactive dose to obtain an adjusted value. The mean cumulative reactive doses at Months 12 and 24 are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: Month 12 and Month 24 (end of treatment) of the OLFUS-VIPES study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 123 | 48
mg
  Month 12: number analyzed (Participants) | 103 | 46
  Month 12 | 1419.6 (1595.92) | 895.9 (1329.14)
  Month 24: number analyzed (Participants) | 83 | 41
  Month 24 | 1751.1 (1962.12) | 758.4 (1176.38)

6. Secondary Outcome: Change From VIPES Baseline in Peanut-Specific Immunoglobulin E (IgE) at Months 6, 12, 18 and 24
Description: The change from the VIPES Baseline in peanut-specific IgE values at Months 6, 12, 18 and 24 of the OLFUS-VIPES study are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: VIPES Baseline to Months 6, 12, 18 and 24 (end of treatment) of the OLFUS-VIPES study
Population: The full analysis set was the intent-to-treat population which consisted of all participants and results are reported for those participants who had the Months 6, 12, 18 and 24 DBPCFC performed.
Measure: Median (Full Range); unit: kilo units per liter
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 123 | 48
kilo units per liter
  VIPES Baseline to Month 6: number analyzed (Participants) | 117 | 48
  VIPES Baseline to Month 6 | 2.150 [-306.00 to 500.12] | 18.900 [-72.37 to 344.79]
  VIPES Baseline to Month 12: number analyzed (Participants) | 104 | 46
  VIPES Baseline to Month 12 | -0.370 [-189.17 to 1168.12] | 4.785 [-447.41 to 233.11]
  VIPES Baseline to Month 18: number analyzed (Participants) | 95 | 43
  VIPES Baseline to Month 18 | -1.870 [-1091.88 to 433.97] | -0.710 [-389.03 to 716.20]
  VIPES Baseline to Month 24: number analyzed (Participants) | 85 | 41
  VIPES Baseline to Month 24 | -3.160 [-381.93 to 861.24] | -10.060 [-384.03 to 332.83]

7. Secondary Outcome: Change From VIPES Baseline in Peanut-Specific Immunoglobulin G Subtype 4 (IgG4) at Months 6, 12, 18 and 24
Description: The change from the VIPES Baseline in peanut-specific IgG4 values at Months 6, 12, 18 and 24 of the OLFUS-VIPES study are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: VIPES Baseline to Months 6, 12, 18 and 24 (end of treatment) of the OLFUS-VIPES study
Population: as for outcome 6
Measure: Median (Full Range); unit: mg/L
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 123 | 48
mg/L
  VIPES Baseline to Month 6: number analyzed (Participants) | 118 | 46
  VIPES Baseline to Month 6 | 1.935 [-6.82 to 28.95] | 0.775 [-0.80 to 8.86]
  VIPES Baseline to Month 12: number analyzed (Participants) | 105 | 44
  VIPES Baseline to Month 12 | 2.890 [-7.06 to 34.80] | 1.510 [-0.61 to 11.93]
  VIPES Baseline to Month 18: number analyzed (Participants) | 95 | 43
  VIPES Baseline to Month 18 | 2.780 [-5.04 to 21.90] | 2.370 [-0.26 to 16.98]
  VIPES Baseline to Month 24: number analyzed (Participants) | 85 | 41
  VIPES Baseline to Month 24 | 2.170 [-5.64 to 27.51] | 1.950 [-0.89 to 15.40]

8. Secondary Outcome: Change From VIPES Baseline in Wheal Diameter During Skin Prick Testing at Months 6, 12, 18 and 24
Description: The change from the VIPES Baseline in the wheal diameter from the undiluted skin prick tests at Months 6, 12, 18 and 24 of the OLFUS-VIPES study are presented according to whether participants received Viaskin Peanut or placebo during the VIPES study.
Time Frame: VIPES Baseline to Months 6, 12, 18 and 24 (end of treatment) in the OLFUS-VIPES study
Population: as for outcome 6
Measure: Median (Full Range); unit: millimeters
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
Number analyzed (Participants) | 123 | 48
millimeters
  VIPES Baseline to Month 6: number analyzed (Participants) | 121 | 48
  VIPES Baseline to Month 6 | -2.30 [-17.0 to 8.5] | -1.50 [-14.0 to 3.5]
  VIPES Baseline to Month 12: number analyzed (Participants) | 106 | 47
  VIPES Baseline to Month 12 | -3.00 [-15.0 to 7.3] | -1.00 [-14.5 to 22.5]
  VIPES Baseline to Month 18: number analyzed (Participants) | 97 | 45
  VIPES Baseline to Month 18 | -3.00 [-27.6 to 8.0] | -1.40 [-14.5 to 10.5]
  VIPES Baseline to Month 24: number analyzed (Participants) | 85 | 43
  VIPES Baseline to Month 24 | -2.00 [-15.0 to 13.0] | -1.50 [-15.0 to 6.5]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from OLFUS-VIPES Baseline up to Month 24. Overall time frame of up to 24 months.
Description: The safety analysis set included all participants who received at least 1 dose of IP during the OLFUS-VIPES study.
Arm/Group | VIPES Initial Treatment Group: All Viaskin Peanut Doses | VIPES Initial Treatment Group: Placebo
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/48
Serious Adverse Events (participants affected / at risk) | 7/123 | 3/48
Other Adverse Events (participants affected / at risk) | 113/123 | 47/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIPES Initial Treatment Group: All Viaskin Peanut Doses (N=123) | VIPES Initial Treatment Group: Placebo (N=48)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIPES Initial Treatment Group: All Viaskin Peanut Doses (N=123) | VIPES Initial Treatment Group: Placebo (N=48)
Conjunctivitis (Eye disorders) | 5 (5) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (10) | 7 (14)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 4 (11)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 2 (2)
Nausea (Gastrointestinal disorders) | 7 (8) | 6 (9)
Vomiting (Gastrointestinal disorders) | 12 (14) | 8 (8)
Application site dermatitis (General disorders) | 9 (12) | 4 (5)
Application site eczema (General disorders) | 14 (18) | 7 (9)
Application site erythema (General disorders) | 69 (238) | 28 (96)
Application site irritation (General disorders) | 5 (6) | 3 (8)
Application site oedema (General disorders) | 7 (13) | 3 (5)
Application site papules (General disorders) | 9 (10) | 7 (7)
Application site pruritus (General disorders) | 57 (194) | 33 (117)
Application site rash (General disorders) | 10 (16) | 8 (16)
Application site swelling (General disorders) | 28 (111) | 20 (67)
Application site urticaria (General disorders) | 9 (27) | 1 (5)
Pyrexia (General disorders) | 18 (32) | 6 (7)
Allergy to animal (Immune system disorders) | 7 (12) | 1 (1)
Food allergy (Immune system disorders) | 14 (37) | 4 (4)
Hypersensitivity (Immune system disorders) | 6 (7) | 4 (7)
Seasonal allergy (Immune system disorders) | 6 (9) | 7 (15)
Ear infection (Infections and infestations) | 3 (5) | 5 (7)
Influenza (Infections and infestations) | 8 (8) | 4 (4)
Nasopharyngitis (Infections and infestations) | 25 (41) | 14 (30)
Pharyngitis streptococcal (Infections and infestations) | 6 (6) | 3 (4)
Rhinitis (Infections and infestations) | 8 (17) | 2 (2)
Sinusitis (Infections and infestations) | 6 (6) | 3 (4)
Upper respiratory tract infection (Infections and infestations) | 17 (37) | 11 (26)
Viral infection (Infections and infestations) | 5 (9) | 3 (4)
Viral upper respiratory tract infection (Infections and infestations) | 3 (6) | 4 (5)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (10) | 2 (2)
Headache (Nervous system disorders) | 25 (80) | 12 (44)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 6 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (28) | 14 (29)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 (26) | 8 (15)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 (19) | 10 (11)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 17 (22) | 9 (12)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 9 (17) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 8 (11) | 4 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (25)
Acne (Skin and subcutaneous tissue disorders) | 6 (7) | 4 (7)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 5 (6) | 4 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 17 (20) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes